CLINICAL TRIAL: NCT05851586
Title: Effectiveness of Physical Therapy Intervention in Pre-Clinical Dental Students
Brief Title: Physical Therapy Intervention in Dental Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joshua Subialka (Other)
Responsible Party: Sponsor-Investigator, Joshua Subialka, Assistant Professor, Associate Investigator, Midwestern University
Organization: Midwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AZ-5178
Record Dates: First submitted 2023-04-20; First posted 2023-05-09 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pain; Strength; Quality of Life
Keywords: Dental students; Supervised exercise; Home exercise program; Strength; Quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised exercise + home exercise program (Experimental): The intervention group (supervised exercise) which will receive supervised strengthening and stretching exercises by a licensed physical therapist in a group setting 2 times per month for 30 minutes each session as well as a home exercise program with general stretching and strengthening exercises for various body parts (focusing on neck, thoracic spine, lumbar spine, shoulder and hand/wrist) that will be identical to the home exercise program only group.
  Interventions: Procedure: Supervised exercise + home exercise program
- Home exercise program only (Active Comparator): The home exercise program only group will be provided with a written home exercise program consisting of general stretching and strengthening exercises for various body parts (focusing on neck, thoracic spine, lumbar spine, shoulder and hand/wrist). The exercise programs will be identical for both the supervised exericse and the home exercise program only groups.
  Interventions: Procedure: Home exercise program only

INTERVENTIONS:
Procedure: Supervised exercise + home exercise program — The supervised exercise + home exercise program group will receive a written home exercise program with general stretching and strengthening exercises for the neck, thoracic spine, lumbar spine, shoulder and hand/wrist. They will also be provided with two supervised exercise sessions per month delivered in a group setting in order to ensure proper performance of the home exercise programs.
  Arms: Supervised exercise + home exercise program
Procedure: Home exercise program only — The home exercise program only group will receive a written home exercise program with general stretching and strengthening exercises for the neck, thoracic spine, lumbar spine, shoulder and hand/wrist, without any supervised guidance on exercise performance.
  Arms: Home exercise program only

SUMMARY:
The main purpose of our study is to assess whether guided strength training and stretching intervention with a written home exercise program is more effective than a home exercise program alone for pre-clinical dental students in improving and preventing pain associated with dental laboratory practice. Secondary aims will be to assess relationships between strength and quality of life measures of an individual and pain levels.

DETAILED DESCRIPTION:
Musculoskeletal (MSK) pain has been identified as a major concern among dental professionals. This can lead to decreased productivity, efficiency and quality of work along with higher costs for the medical system. The body region that is affected the most is the neck, followed by the back and shoulders.

Ergonomic assessments and interventions can identify the areas of concern with workplace set up, however, training the muscles to adapt to abnormal postures may be an effective way of increasing the resilience of the MSK system while decreasing MSK pain as well. Specifically, strength training and stretching has been well researched as a way to prevent and improve pain for neck pain, low back pain and shoulder pain. Physical therapists are well trained in prevention and treatment of injuries, including a wealth of knowledge regarding strength training and stretching for specific regions. The main purpose of our study is to assess whether guided strength

Thus, the main purpose of our study is to assess whether guided strength training and stretching intervention with a written home exercise program is more effective than a home exercise program alone for pre-clinical dental students in improving and preventing pain associated with dental laboratory practice. The secondary aim will be to assess the relationships between strength and quality of life measures of an individual and pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18+
* Current 2nd year university dental students

Exclusion Criteria:

* Any type of musculoskeletal surgery in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline
  PROMIS® is a publicly available system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. This will be measured via electronic survey.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Intervention conclusion (7 months)
  PROMIS® is a publicly available system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. This will be measured via electronic survey.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 11 months
  PROMIS® is a publicly available system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. This will be measured via electronic survey.
Pain Intensity | Baseline
  Visual analog scale (0-10 rating)
Pain Intensity | Intervention conclusion (7 months)
  Visual analog scale (0-10 rating)
Pain Intensity | 11 months
  Visual analog scale (0-10 rating)

SECONDARY OUTCOMES:
Pec Minor Length Test | Baseline, intervention conclusion (7 months), and 4 month follow up prior to beginning clinical rotations.
  Supine measurement in centimeters from table
Pec Minor Length Test | Intervention conclusion (7 months)
  Supine measurement in centimeters from table
Pec Minor Length Test | 11 months
  Supine measurement in centimeters from table
Middle Trapezius Manual Muscle Test | Baseline
  Patient prone with arms abducted to 90 degrees and externally rotated, resisting horizontal adduction. Measured in lbs or Newtons using a handheld dynamometer.
Middle Trapezius Manual Muscle Test | Intervention conclusion (7 months)
  Patient prone with arms abducted to 90 degrees and externally rotated, resisting horizontal adduction. Measured in lbs or Newtons using a handheld dynamometer.
Middle Trapezius Manual Muscle Test | 11 months
  Patient prone with arms abducted to 90 degrees and externally rotated, resisting horizontal adduction. Measured in lbs or Newtons using a handheld dynamometer.
Lower Trapezius Manual Muscle Test | Baseline
  Patient prone with arms abducted 120 degrees and externally rotated, resisting downward force. Measured in lbs or Newtons using a handheld dynamometer.
Lower Trapezius Manual Muscle Test | Intervention conclusion (7 months)
  Patient prone with arms abducted 120 degrees and externally rotated, resisting downward force. Measured in lbs or Newtons using a handheld dynamometer.
Lower Trapezius Manual Muscle Test | 11 months
  Patient prone with arms abducted 120 degrees and externally rotated, resisting downward force. Measured in lbs or Newtons using a handheld dynamometer.
Cervical Flexor Endurance Test | Baseline
  Patient in supine will be asked to tuck the chin and lift their head maintaining the chin tuck. Measured in seconds for as long as they can maintain appropriate quality of movement.
Cervical Flexor Endurance Test | Intervention conclusion (7 months)
  Patient in supine will be asked to tuck the chin and lift their head maintaining the chin tuck. Measured in seconds for as long as they can maintain appropriate quality of movement.
Cervical Flexor Endurance Test | 11 months
  Patient in supine will be asked to tuck the chin and lift their head maintaining the chin tuck. Measured in seconds for as long as they can maintain appropriate quality of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Lacey Frankland, DPT, Principal Investigator — Midwestern University
Locations (1):
- Midwestern University, Glendale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No